CLINICAL TRIAL: NCT06536361
Title: The Effect of a Virtual Reality-Based Learning Tool on Nursing Students' Knowledge and Skills in Thorax and Lung Physical Examination
Brief Title: Impact of a VR-Based Learning Tool on Nursing Students' Skills in Thorax and Lung Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Nurcan Çalışkan, Professor of Nursing, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023-915; 2024-9040 (Other Grant/Funding Number: GAZI UNIVERSITY RESEARCH PROJECTS UNIT (BAP))
Record Dates: First submitted 2024-07-23; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Nurse's Role; Nurse-Patient Relations; Exanimation
Keywords: Physical Examination; Virtual Reality; Nursing Education; Thorax; Lung; Simulation Training; Educational Technology
MeSH Terms: conditions — Coma

STUDY DESIGN:
Intervention Model Description: This study is a single-blind, pre-test-post-test, parallel group randomized controlled trial. Participants will first receive theoretical training, followed by demonstration videos one week later. Skills training in the simulation lab will be conducted two weeks after the theoretical training. At the semester's end, participants will be assigned to groups based on gender and course achievement scores. Two weeks before the intervention, pre-reading materials and demonstration videos for thorax and lung physical examination will be distributed. Knowledge and skill levels will be assessed seven days before the intervention. The control group will receive skills training in small groups using a manual and practice on each other. The experimental group will use a VR-based learning tool for training. Final assessments will take place seven days after the intervention, with experimental group students providing feedback on the VR tool's usability.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding: Participant blinding was implemented in the study. Participants were recruited without being informed of their group assignments, and different teaching techniques were applied to each group sequentially. The participants' skills were assessed by a field expert who was unaware of their group allocation. During the data collection phase, data were entered into the system by an individual other than the researcher and subsequently shared with an independent statistical expert without revealing group assignments. This expert conducted the data analysis without knowledge of which group was assigned to the experimental condition and which to the control condition. Blinding of outcome assessment was ensured, thereby minimizing bias. The blinding of evaluators, participants, and statisticians was employed to control for detection and statistical biases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality-Based Learning Tool Group (Experimental): At the beginning of the study, all participants will receive theoretical training. One week later, they will review the topic through thorax and lung physical examination videos. Two weeks after theoretical training, participants will undergo skills training in the simulation laboratory. At the semester's end, participants taking the final exam will be grouped based on gender and course success scores. Two weeks before the intervention, pre-reading materials and demonstration videos will be distributed. Knowledge and skill levels will be assessed seven days prior to the intervention. The experimental group will receive training using a VR-based learning tool. Final assessments will occur seven days post-intervention. Feedback on the VR tool from the experimental group will be collected using a student opinion form after the final skills assessment.
  Interventions: Other: Virtual Reality-Based Learning Tool
- Traditional Small Group Training (Active Comparator): At the beginning of the study, all participants will receive theoretical training. One week later, the topic will be reviewed through thorax and lung physical examination videos. Two weeks after the theoretical training, participants will undergo skills training in the simulation laboratory. At the end of the semester, participants will take a final exam and be assigned to research groups based on their gender and course success scores. Two weeks prior to the implementation, pre-reading materials and thorax and lung physical examination videos will be distributed. Knowledge and skill levels will be assessed seven days before the implementation. Students in the control group will receive training in small groups in the skills laboratory, using the thorax and lung physical examination skills control form. Following the training, all participants will practice on each other. Final knowledge and skills assessments will be conducted seven days after the intervention
  Interventions: Other: Traditional Small Group Training

INTERVENTIONS:
Other: Virtual Reality-Based Learning Tool — The intervention involves the use of a virtual reality-based learning tool to teach thorax and lung physical examination skills. The tool uses Oculus Meta Quest 3 VR headset to provide immersive simulation experiences. The VR tool includes high-quality graphics and interactive scenarios to facilitate skill development.
  Arms: Virtual Reality-Based Learning Tool Group
Other: Traditional Small Group Training — The intervention involves traditional small group training conducted in the Nursing Principles Skills Laboratory. This training includes hands-on practice with physical examination techniques using simulation mannequins and feedback from instructors. The approach is designed to provide practical experience without the use of virtual reality technology.
  Arms: Traditional Small Group Training

SUMMARY:
Short Title: Impact of VR-Based Learning Tools on Nursing Students' Thoracic and Lung Examination Skills

Short Summary: This study evaluates the impact of a virtual reality (VR) based learning tool on nursing students' knowledge and skills in thoracic and lung physical examinations. Designed as a single-blind, pre-test-post-test, control group, parallel-group randomized controlled trial in accordance with SPIRIT 2013 guidelines, the study was conducted with 82 second-year nursing students from Gazi University, comprising 41 students in the experimental group and 41 in the control group. Initially, participants were informed about the study and received theoretical training during the first week. The second week included a review through demonstration videos, while the third week involved hands-on practice using high-fidelity simulators in a skills lab for auscultation and physical examination. The final exam was administered in the fifth week. Participants meeting eligibility criteria were stratified by gender and academic performance, then randomly assigned to groups by an independent statistician. Pre-reading materials were distributed one week before the intervention, followed by an evaluation of knowledge and skill levels. The experimental group underwent VR-based training, whereas the control group received traditional instruction. Final assessments of knowledge and skills were conducted one week post-training. Data collection included demographic forms, knowledge tests, skill assessments, and student feedback. Blinding was applied to evaluators, participants, and statisticians to minimize bias. Data analysis will employ statistical software, utilizing parametric tests for normally distributed data and non-parametric tests for non-normally distributed data.

Study Type: Interventional Study Design: Single-blind, pre-test-post-test, control group, parallel-group randomized controlled trial.

Primary Outcomes:

Knowledge and skill levels (Measured by knowledge tests and skill assessment forms)

Secondary Outcomes:

Participant feedback on the VR-based learning tool (Assessed through student feedback forms)

Eligibility Criteria:

Second-year nursing students at Gazi University enrolled in the "Health Assessment" course, who have passed with at least a CC grade, have an academic success score between 2.00 and 4.00, are willing to participate, and do not have visual impairments affecting depth perception (e.g., amblyopia, anisometropia, strabismus).

DETAILED DESCRIPTION:
Purpose of the Research: The study was designed to determine the effect of a virtual reality (VR)-based learning tool for thorax and lung physical examination on nursing students' knowledge and skills related to thorax and lung physical examination.

Hypotheses of the Study:

Hypothesis 0-1: There is no significant difference in the knowledge of thorax and lung physical examination between students in the experimental group using the VR-based learning tool and students in the control group receiving small group instruction.

Hypothesis 1-1: There is a significant difference in the knowledge of thorax and lung physical examination between students in the experimental group using the VR-based learning tool and students in the control group receiving small group instruction.

Hypothesis 0-2: There is no significant difference in the skills related to thorax and lung physical examination between students in the experimental group using the VR-based learning tool and students in the control group receiving small group instruction.

Hypothesis 1-2: There is a significant difference in the skills related to thorax and lung physical examination between students in the experimental group using the VR-based learning tool and students in the control group receiving small group instruction.

Research Question: What are the opinions of students in the experimental group regarding the use of the VR-based thorax and lung physical examination learning tool? Variables of the Study

Independent Variables:

Training Method: Small group instruction for the control group; VR-based thorax and lung physical examination learning tool for the experimental group.

Dependent Variables:

Knowledge Level: Knowledge as measured by pre-test and post-test results. Skill Level: Skill level assessed by pre-skill and post-skill measurements.

Control Variables:

Participants' gender. Participants' course achievement scores. Materials and Method Type of Research: This study was designed as a single-blind, pretest-posttest, control group, parallel-group randomized controlled trial. The study was conducted in accordance with the SPIRIT 2013 guidelines. To minimize bias, the study protocol will be registered in the Clinical Trials registration system.

Location Characteristics and Time of the Research The study was conducted with students enrolled in the elective course "Health Assessment" (HEM 205) at Gazi University Faculty of Nursing during the 2023-2024 academic year. This two-credit elective course covers physical examination methods and techniques both theoretically and practically. Theoretical instruction occurs in classrooms, while practical training is provided in skills and simulation laboratories by field experts.

Population and Sample of the Study: The study population comprised second-year nursing students who had successfully completed their first year and were enrolled in the second year during the 2023-2024 academic year, and who selected the "Health Assessment" elective course (HEM 205) for the first time. The sample size for the study was calculated using GPower version 3.1.9.7 software. The sample size calculation in GPower utilized a t-test to assess the mean difference between two independent groups, with a priori values of α = 0.05, power = 0.90, and a large effect size (f = 0.80 Cohen's d). Based on the statistical analysis, a total sample of 68 participants was determined, with 34 assigned to the control group and 34 to the experimental group. In experimental research, it is critical to keep participant loss below 20% to minimize bias, and increasing the sample size helps control for potential bias due to attrition. To address potential losses, the study aimed to include 41 participants in each group, resulting in a total sample size of 82 participants.

Randomization: The randomization process was conducted in accordance with the CONSORT 2017 guidelines. An independent statistician stratified participants based on their achievement scores in the "Health Assessment" course and their gender. Female students with achievement scores between 2.00-3.00 (CC, CB, BB) were placed in the first stratum, while those with scores between 3.01-4.00 (BA, AA) were placed in the second stratum. Male students with achievement scores between 2.00-3.00 (CC, CB, BB) were assigned to the third stratum, and those with scores between 3.01-4.00 (BA, AA) were assigned to the fourth stratum. The statistician then performed simple randomization within each stratum using Excel software, resulting in random assignment of 41 students to the experimental group and 41 students to the control group.

Data Collection Tools Descriptive Characteristics Form: Developed by the researcher based on the literature, this form consists of fourteen questions. It includes eight questions regarding the demographic characteristics of the participants, one question concerning their eye health, one question about their willingness to choose the nursing profession, and four questions related to their technological attitudes.

Thorax and Lung Physical Examination Knowledge Test: Created by the researcher in alignment with the subject scope and learning objectives of the theoretical course on thorax and lung physical examination. This test comprises 20 questions with five options each, assessing knowledge necessary for performing thorax and lung physical examinations. Each question is scored out of 5 points, with higher scores indicating greater knowledge levels.

Thorax and Lung Physical Examination Skill Control Form: Designed to assess the initial and final skill levels of the students. This form, developed in accordance with the literature, includes a total of 48 procedural steps. Scores range from 0 to 96, with higher scores reflecting higher skill levels.

Student Opinion Form: Prepared by the researcher following relevant literature to gauge student opinions on the VR-based learning tool. This form has two sections. The first section, based on the technology acceptance model and literature review, consists of 29 items evaluating the ease of use (14 items) and perceived usefulness (15 items) of the VR tool. The second section contains six open-ended questions about the VR-based thorax and lung physical examination learning tool.

Content Validity Analysis Content validity was assessed by consulting 13 experts in physical examination methods and innovative digital education. They rated the forms on a 4-point Likert scale (4: Very appropriate, 3: Appropriate with minor adjustments, 2: Appropriate with major adjustments, 1: Not appropriate) regarding purpose, objectives, language, and expression. Expert opinions were analyzed using Davis's technique to calculate the content validity index, and agreement was tested with Kendall's W.

Designing a VR-Based Learning Tool

In designing the VR-based thorax and lung physical examination learning tool, the "Healthcare Implementation Standards of Best Practice Simulation Design" guide provided by the International Nursing Association for Clinical Simulation and Learning (INACSL) was used as the foundation. The design process was structured as follows:

Analysis Phase: The researcher completed training necessary for effective simulation design. Existing training methods of the target group were evaluated through SWOT analysis. The objectives of the learning tool were defined using SMART analysis.

Design Phase: The relevant literature was reviewed to determine the simulation method and scenario to be employed. The interaction methods within the VR learning tool and the scenario outline were developed.

Development Phase: High-quality graphics, models, and interaction methods were utilized to enhance the realism of the learning tool. Facilitative approaches were planned to support the participants' learning process.

Implementation Phase: Materials to guide the learning tool were prepared. The PEARLS method was employed to evaluate the learning tool following the simulation implementation. The tool's applicability and usability were assessed by participants, and necessary adjustments were made based on the feedback received from the pre-application.

Pre-Application: To evaluate the VR-based learning tool and data collection instruments, a pre-application was conducted with third-year students at Gazi University Faculty of Nursing who had previously completed the elective course "Health Assessment" (coded HEM 205). This pre-application assessed the clarity of the data collection tools in terms of language and expression, as well as the usability of the VR-based learning tool.

Application:

In the first week of the study, all participants underwent theoretical training. The second week included a review of the topic through demonstration videos, and skills training in the simulation laboratory was conducted in the third week. By the fifth week, all participants completed the final exam. Participants were then stratified and assigned to research groups based on their gender and course achievement scores.

The VR-based thorax and lung physical examination learning tool for the experimental group was designed and developed over a period of five months. During this time, all necessary preparations were completed. Pre-reading materials and demonstration videos were distributed to the participants. Seven days following the distribution of these materials, initial knowledge and skill assessments were conducted.

Practical training took place seven days after the initial assessments. The control group received 55 minutes of training in groups of 8, which included 7 minutes for an overview of the training purpose and content, 40 minutes for hands-on practice (5 minutes per student), and 8 minutes for feedback. The experimental group used the VR-based tool for 35 minutes, which comprised 7 minutes for an introduction to the Oculus Meta Quest 3, 20 minutes for skill practice on a virtual patient, and 8 minutes for a debriefing session.

Final knowledge and skill assessments were carried out seven days post-intervention. The experimental group participants completed the Student Opinion Form to provide feedback on the usability and applicability of the VR-based tool. Additionally, they received further training with the VR-based tool after the completion of all measurements and evaluations.

Analysis: Data will be analyzed using a computer program. The normal distribution of variables will be assessed through histograms, coefficient of variation, skewness, kurtosis, Kolmogorov-Smirnov, and Shapiro-Wilk tests (p<0.05). Descriptive statistics (number, percentage, mean, standard deviation) and Chi-square tests will be used. Parametric tests will be applied to normally distributed data, while non-parametric tests will be applied to non-normally distributed data. An independent sample t-test will be used for comparisons between two independent groups, ANOVA with Bonferroni correction for comparisons among more than two groups, and analysis of variance for repeated measures. For non-normally distributed data, Mann-Whitney U and Kruskal-Wallis H tests with Bonferroni correction will be applied. Randomization balance will be maintained using Intention-to-Treat (ITT) analysis.

Limitations of the Study: This study was conducted exclusively with second-year students enrolled at the Faculty of Nursing of a university in Turkey. This limitation affects the generalizability of the research findings, as the results may not be directly applicable to other student populations or educational settings.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study.
* Ability to understand and speak Turkish,
* Absence of eye conditions affecting depth perception, such as amblyopia (lazy eye), anisometropia (different refractive errors in each eye), and strabismus (squint). (Self- report is accepted.),
* Academic performance score between 2.00 and 4.00.,
* Enrollment in the HEM 205 "Health Assessment" course for the first time in the Fall Semester of the 2023-2024 academic year,
* Obtaining at least a CC grade in the HEM 205 "Health Assessment" course.

Exclusion Criteria:

* The participant expresses a desire to withdraw from the study,
* Failure to attend the theoretical course on thorax and lung physical examination,
* Failure to watch the demonstration videos for thorax and lung physical examination,
* Failure to participate in laboratory sessions,
* Failure to complete data collection forms (Student Identification Form, Knowledge Test, and Student Opinion Form) or incomplete completion of these forms,
* Failure to participate in small group training sessions,
* Failure to use the virtual reality-based thorax and lung physical examination training tool,
* Failure to participate in any stage of the skill assessment is a criterion for exclusion from the study.

Criteria for Exclusion from the Study:

* The student is a graduate of a high school, associate degree, or undergraduate program in a health-related field.
* The student is retaking the course HEM 205 "Health Assessment."
* These are the criteria for exclusion from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Knowledge Level of Thorax and Lung Physical Examination | Knowledge levels will be evaluated seven days prior to the intervention (pre-test) and seven days following the intervention (post-test).
  This outcome measure assesses nursing students' theoretical understanding of thorax and lung physical examination procedures through a knowledge test. Scores range from 0 to 100, with higher scores indicating enhanced theoretical knowledge. The unit of measure is the score, which can range from 0 to 100 points.
Skill Level in Thorax and Lung Physical Examination | Skill levels will be assessed seven days before the intervention (pre-test) and seven days after the intervention (post-test).
  This measure evaluates the practical application of thorax and lung physical examination techniques using a skill control form. Scores range from 0 to 96, with higher scores reflecting improved practical skills. The unit of measure is the score, which can range from 0 to 96 points.

SECONDARY OUTCOMES:
Usability Feedback on the VR Tool | Feedback will be collected immediately after the final skills measurement.
  This measure collects feedback from the experimental group regarding the usability of the VR-based learning tool. Feedback will be gathered using a student opinion form featuring a 5-point Likert scale. The unit of measure is the Likert scale rating, which ranges from 1 to 5 points.
Applicability Feedback on the VR Tool | Feedback will be collected immediately after the final skills measurement.
  This measure gathers students' opinions on the applicability of the VR-based learning tool, including detailed feedback through open-ended questions. The same student opinion form used for usability feedback will be employed. The unit of measure includes both the Likert scale rating (1 to 5 points) and qualitative feedback.
Student Opinions on the VR-Based Learning Tool | Feedback will be collected immediately after the final skills measurement.
  This measure collects detailed feedback from students in the experimental group regarding the VR-based learning tool. Feedback is gathered through a section consisting of six open-ended questions. These questions are designed to elicit comprehensive insights into students' experiences, suggestions, and overall perceptions of the VR tool. The unit of measure includes qualitative data from the responses to the open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan Çalışkan, Prof.Dr., Study Director — Gazi University Nursing Faculty
Locations (1):
- Gazi University Nursing Faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Padilha JM, Machado PP, Ribeiro A, Ramos J, Costa P. Clinical Virtual Simulation in Nursing Education: Randomized Controlled Trial. J Med Internet Res. 2019 Mar 18;21(3):e11529. doi: 10.2196/11529. PMID 30882355
- [Background] Bayram SB, Caliskan N. Effect of a game-based virtual reality phone application on tracheostomy care education for nursing students: A randomized controlled trial. Nurse Educ Today. 2019 Aug;79:25-31. doi: 10.1016/j.nedt.2019.05.010. Epub 2019 May 9. PMID 31102793
- [Background] Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P; CONSORT NPT Group. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 2017 Jul 4;167(1):40-47. doi: 10.7326/M17-0046. Epub 2017 Jun 20. PMID 28630973
- [Background] Akın, B. ve Koçoğlu, D. Randomize Kontrollü Deneyler. Hacettepe Üniversitesi Hemşirelik Fakültesi Dergisi. 2017 4(1): 73-92.
- [Background] Han SG, Kim YD, Kong TY, Cho J. Virtual reality-based neurological examination teaching tool(VRNET) versus standardized patient in teaching neurological examinations for the medical students: a randomized, single-blind study. BMC Med Educ. 2021 Sep 15;21(1):493. doi: 10.1186/s12909-021-02920-4. PMID 34526004
- [Background] Yang TY, Huang CH, An C, Weng LC. Construction and evaluation of a 360 degrees panoramic video on the physical examination of nursing students. Nurse Educ Pract. 2022 Aug;63:103372. doi: 10.1016/j.nepr.2022.103372. Epub 2022 May 24. PMID 35644047
- [Background] Cheung VYT, Tang YM, Chan KKL. Medical students' perception of the application of a virtual reality training model to acquire vaginal examination skills. Int J Gynaecol Obstet. 2023 Jun;161(3):827-832. doi: 10.1002/ijgo.14670. Epub 2023 Jan 31. PMID 36637241
- [Background] Hogan-Quigley, B., Palm, M. L., Bickley, L. S. 2012. Bates' nursing guide to physical examination and history taking. Philadelphia, PA: Lippincott Williams & Wilkins.
- [Background] Hogan-Quigley, B., Palm, M. L., Bickley, L. S. 2017. ''Bates' Nursing Guide to Physical Examination and History Taking. 2nd edtion'', Philadelphia: Wolters Kluwer, pp 292-299.
- [Background] Weber, J. R., Kelley, J. H. 2014. ''Assessing Thorax and Lung in Health Assessment in Nursing''. 5th edition Lippincott Williams & Wilkins. pp 369-390
- [Background] Chaplen, R. 2019. ''Thorax and Lung Assessment içinde Nursing health assessment: A best practice approach''. Editör Jensen, S. 3rd Edition, Lippincott Williams & Wilkins. pp 668-682
- [Background] Görgülü, R. S. 2014. Hemşireler için fiziksel muayene yöntemleri. 1. Baskı (pp. 79-94). İstanbul Medikal Yayıncılık.
- [Background] Benzaghta, M. A., Elwalda, A., Mousa, M., Erkan, I., & Rahman, M. (2021). SWOT analysis applications: An integrative literature review. Journal of Global Business Insights, 6(1), 55-73. https://doi.org/10.5038/2640-6489.6.1.1148
- [Background] May, R., Tyndall, I., McTiernan, A., Roderique-Davies, G., & McLoughlin, S. (2022). The impact of the SMART program on cognitive and academic skills: a systematic review and meta-analysis. British Journal of Educational Technology, 53(5), 1244-1261. Advance online publication. https://doi.org/10.1111/bjet.13192
- [Background] Eppich W, Cheng A. Promoting Excellence and Reflective Learning in Simulation (PEARLS): development and rationale for a blended approach to health care simulation debriefing. Simul Healthc. 2015 Apr;10(2):106-15. doi: 10.1097/SIH.0000000000000072. PMID 25710312
- [Background] INACSL Standards Committee. (2021). Healthcare Simulation Standards of Best PracticeTM Simulation Design. Clinical Simulation in Nursing, 58, 14-21
- [Background] Pereira D, Gomes P, Faria S, Cruz-Correia R, Coimbra M. Teaching cardiopulmonary auscultation in workshops using a virtual patient simulation technology - A pilot study. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:3019-3022. doi: 10.1109/EMBC.2016.7591365. PMID 28268948